CLINICAL TRIAL: NCT00438620
Title: A Pilot Study to Explore the Role of Physical Activity as a Quality of Life Intervention in Advanced Cancer Patients
Brief Title: The Feasibility of Physical Activity in Advanced Cancer Patients
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PS-08-0054
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Home-based physical activity program — the role of physical activity as a Quality of Life intervention

SUMMARY:
Physical activity has been shown to have a positive effect on several quality of life outcomes in cancer patients, but few existing studies have focused on the end stages of cancer. The aim of this pilot study is to test the feasibility of a physical activity intervention in advanced cancer patients, from which data can be used to design a randomized controlled trial if results are encouraging.

DETAILED DESCRIPTION:
Background Information Cancer is one of the leading causes of mortality and morbidity worldwide[1]. The resultant morbidities of cancer and its treatment are manifold; common physiologic symptoms include pain, muscle weakness and fatigue, whereas common psychological symptoms include depression, anxiety and poor sense of well-being. As methods of cancer detection and treatment improve, survival is prolonged and the lifetime burden of these adverse effects increases[2]. Addressing these issues is critical towards maximizing quality of life, a multidimensional construct encompassing all physical and psychosocial factors[3].

Physical activity is one potential strategy for ameliorating quality of life in all phases of cancer and its treatment [4]. Increasing evidence indicates a role for physical activity in improving several aspects of physical and psychological well-being that may contribute to quality of life in cancer patients, including muscle strength, functional capacity, mood and self-esteem[5]. Not only does physical activity have proven benefits in terms of physical performance and fatigue in cancer survivors, it may improve the capacity for basic activities of daily living such that functional independence can be maintained as long as possible[6]. Although this has been demonstrated for early stage cancer survivors, there is limited evidence for the use of physical activity in the palliation of patients with actively progressive, advanced incurable cancer[7]. A few studies of exercise in advanced metastatic cancer patients have demonstrated benefits in quality of life outcomes, however small sample sizes have limited their generalizability to the larger end-stage cancer population[8-12]. There exists a critical need to more specifically identify exercise programmes targeted to advanced cancer patients' needs, interests and preferences[13].

Purpose The purpose of this pilot study is to explore the physical activity preferences and interests of actively progressive, advanced incurable cancer patients and to determine if there is any association between physical activity and quality of life in this population. The ultimate aim of this study is to provide preliminary data on which a subsequent intervention trial can be based if encouraging results are obtained.

Objectives

1. To describe advanced cancer patient's attitudes towards physical activity, self-efficacy for physical activity and programming preferences.
2. To examine the relationship between quality of life, medical and demographic variables, and physical activity in advanced cancer patients.
3. To identify which advanced cancer populations would be willing and able to participate in a physical activity intervention.

Study Design This pilot study will be cross-sectional in design, using a survey questionnaire combining both closed and open-ended questions. After written consent is obtained, the investigator will administer the survey questionnaire via face-to-face interview with the patient at a time and location that is mutually convenient for both parties. The survey questionnaire will be a one-time assessment, with anticipated duration of 45 minutes for completion. The survey questionnaire will be developed based on combination of validated physical activity and quality of life questionnaires, including the McGill Quality of Life Questionnaire[14], the Edmonton Symptom Assessment Scale[15], and the Late-Life Function and Disability Instrument[16]. Exercise program preferences and Theory of Planned Behavior constructs will be assessed using items taken from previous research assessing physical activity in cancer survivors[17-19]. Medical and demographic information will be collected using self-report measures and via medical chart review. Date of death will be determined from the cancer registry.

Inclusion Criteria

1. 18 years of age or older
2. Be able to understand, provide written informed consent in, and speak English
3. Cognitive ability to participate (defined as a normal Folstein's Mini Mental Status Score for patient's age and education level[20])
4. Diagnosis of advanced cancer (defined as progressive, incurable, locally recurrent or metastatic disease)
5. Approval of treating physician Exclusion Criteria

1. Any absolute contraindications to exercise (including acute MI within 2 days, symptomatic/severe aortic stenosis, decompensated heart failure, symptomatic/hemodynamically significant cardiac arrhythmias, unstable angina not previously stabilized by medical therapy, acute aortic dissection, acute myocarditis/pericarditis, acute pulmonary embolus/infarction) 2. Palliative Performance Status level of 30% or less[21] 3. Any patient who, in the opinion of the treating physician, is within the last days to hours of life Recruitment Patients diagnosed with advanced cancer (defined as progressive, incurable, locally recurrent or metastatic disease) will be recruited from the Cross Cancer Institute and the Capital Health Regional Palliative Home Care Program. Eligible patients will be identified by case managers in the Capital Health Regional Palliative Home Care Program, and study information will be included in the ethics-approved Pain and Symptom & Palliative Care Research Group studies brochure distributed to outpatients at the Cross Cancer Institute by the research nurse or study coordinator. Patient contact will be made by telephone outside of the Cross Cancer Institute thereafter. Patients who accept the invitation to participate will provide written consent prior to commencing the study.

Statistical Analysis To detect a change of 0.5 standard deviations (a medium effect size) in the various outcomes (quality of life, physical activity) with a power of 80% and a two-tailed alpha value of <0.05, we need 29 participants. Based on previous study sampling of the Cross Cancer Institute and Capital Health Regional Palliative Home Care by the Pain & Symptom and Palliative Care Research Group, 30 patients could be expected to be recruited over a nine month period given frailty and end-of-life symptom limitations. The study will commence with the enrollment of the first subject, subsequent subjects will be recruited on an ongoing basis. Initial analysis will provide complete descriptive information on the demographic and medical profile of the study participants. Primary analysis will use multiple regression to explore the relationship between demographic/medical characteristics, physical function and quality of life variables.

Data Safety Monitoring Committee Ethical and scientific approval will be obtained from the local Institutional Review Boards affiliated with the Cross Cancer Institute and Capital Health Regional Palliative Home Care prior to study commencement. All serious adverse events will be reported to the local IRBs as well as each participant's treating physician. The project coordinator, under the supervision of the principal investigator, will be responsible for reporting any serious adverse events. The local IRBs will oversee the validity and integrity of data by conducting periodic audits of study records.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to understand, provide written consent in and speak English
* cognitive ability to participate
* clinician-estimated life expectancy between 3 and 12 months
* approval of treating physician

Exclusion Criteria:

* any absolute contraindications to physical activity
* palliative performance scale level of 30% of less
* any patient within the last days to hour of life

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Cancer Patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, PhD, Study Chair — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Lowe SS, Watanabe SM, Baracos VE, Courneya KS. Home-based functional walking program for advanced cancer patients receiving palliative care: a case series. BMC Palliat Care. 2013 May 11;12:22. doi: 10.1186/1472-684X-12-22. eCollection 2013. PMID 23663868